CLINICAL TRIAL: NCT05933746
Title: The Impact of a Remote, Brief, Sleep Hygiene Intervention on Undergraduate Students' Sleep and Stress: A Randomized, Controlled Trial
Brief Title: Sleep Hygiene Intervention on Undergraduate Students' Sleep and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark A. Lumley, Distinguished Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-21-10-4095
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Stress, Emotional; Sleep Disturbance
MeSH Terms: conditions — Stress, Psychological; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Condition assignment is done automatically, on-line, to two active experiences. Follow-up assessment is done automatically (on-line measure completion).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Hygiene Intervention (Experimental): 1-hour, on-line set of three modules pertaining to various sleep hygiene behaviors
  Interventions: Behavioral: Sleep Hygiene Intervention
- Non-behavioral Sleep Education (Placebo Comparator): active, matched placebo condition that controls for engagement and rationale
  Interventions: Behavioral: Non-behavioral Sleep Education

INTERVENTIONS:
Behavioral: Sleep Hygiene Intervention — This 1-hour on-line intervention presents three sleep hygiene modules, selected randomly from among these six: establishing a bedtime routine, optimizing sleep environment, implementing a sleep schedule, bedtime relaxation, nutrition choices, and exercise habits.
  Arms: Sleep Hygiene Intervention
Behavioral: Non-behavioral Sleep Education — 1-hour on-line set of three modules that cover non-skill (non-hygiene) educational topics (sleep research, sleep stages, dreams). This control condition equates for engagement rationale.
  Arms: Non-behavioral Sleep Education

SUMMARY:
Poor sleep is common among college students and likely contributes to stress. The investigators developed a brief, remotely-delivered intervention and tested whether it improves sleep hygiene and reduced sleep disturbance and stress among undergraduates.

DETAILED DESCRIPTION:
Poor sleep is common among college students and likely contributes to stress. The investigators developed a brief, remotely-delivered sleep hygiene intervention, which is delivered via the internet, and tested in a randomized controlled trial, whether it improves sleep hygiene and reduced sleep disturbance and stress in a sample of undergraduates who report wanting to improve their sleep. This study compares the novel sleep hygiene intervention to an active, matched control condition--sleep education. Baseline and 2-week follow-up questionnaires assess sleep hygiene, sleep disturbance, and stress. ANCOVAs will compare conditions at follow-up, and mediation tests will explore whether the intervention reduced stress through improved sleep.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students at Wayne State University
* Self-reported desire to improve their sleep

Exclusion Criteria:

* Graduate students / professional students

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Sleep disturbance short-form b | Change from baseline to 2-week follow-up
  8-item measure assesses sleep disturbances over last 7 days (range: 8 to 40; higher scores = more sleep disturbance)

SECONDARY OUTCOMES:
Perceived Stress Scale | Change from baseline to 2-week follow-up
  10-item measure of perceived stress over past 7 days (range 0 to 40; higher scores = more perceived stress)
Sleep Hygiene Inventory | Change from baseline to 2-week follow-up
  13-item measure of maladaptive sleep hygiene behaviors over last 7 days (range: 13-65; higher scores = worse hygiene)

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data set, upon reasonable request